CLINICAL TRIAL: NCT04643691
Title: Benefit of Treatment With Losartan and Spironolactone on the Regulation of the Renin-angiotensin System in the Prognosis of Patients Infected With COVID-19 and Suffering From Acute Respiratory Distress Syndrome
Brief Title: Losartan and Spironolactone Treatment for ICU Patients With COVID-19 Suffering From ARDS
Acronym: COVIDANCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to an Urgent Security Measure
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-24; 2020-001766-11 (EudraCT Number)
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; ARDS
Keywords: COVID-19; ARDS
MeSH Terms: conditions — COVID-19 | interventions — Losartan; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- losartan / spironolactone (Experimental): Losartan 50 mg and Spironolactone 25 mg pillules oral use
  Interventions: Drug: Losartan 50 mg and Spironolactone 25 mg pillules oral use
- usual care (No Intervention): Usual care of COVID-19 infection in intensive care

INTERVENTIONS:
Drug: Losartan 50 mg and Spironolactone 25 mg pillules oral use — Losartan 50 mg and Spironolactone 25 mg pillules oral use during 10 days
  Arms: losartan / spironolactone

SUMMARY:
Coronavirus disease (COVID-19) is a current pandemic infection caused by an RNA virus called Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2). Severe forms of COVID-19 are most often responsible for isolated respiratory failure in the form of acute respiratory distress syndrome (ARDS), which accounts for most of the mortality. Angiotensin converting enzyme 2 (ACE2) has been shown to be a co-receptor for the entry of SARS-CoV-2 into cells and is likely to play a prolonged role in the pathogenesis of COVID-19. ACE2 and angiotensin (1-7) have been shown to be protective in a number of different lung lesion models. In a mouse model of acidic lung injury, negative regulation of ACE2 by COVID, the SARS virus responsible for the 2003 SARS outbreak, worsened the lung injury which was improved by treatment with ARBs.

We believe that blocking the first RAS pathway at the end of the chain on the AT1r angiotensin 2 receptor may prevent the initiation of this chain reaction and limit decompensation secondary to the disruption of the equilibrium of the renin-angiotensin system. We have several molecules that block the AT1r angiotensin-2 receptor (ARBs) as well as a molecule that blocks the secretion of aldosterone (spironolactone). The main objective is to demonstrate the value of losartan and spironolactone therapy in the regulation of the renin-angiotensin system in improving the prognosis of patients infected with COVID-19 and suffering from acute respiratory distress syndrome.

This is a prospective, multicenter, randomized, open-label, controlled, therapeutic trial studying two parallel groups. The population included in this study is any major patient in acute respiratory distress hospitalized in intensive care requiring oxygen support of at least 6L/min and suffering from a PCR-confirmed SARS-cov2 infection. The control group will benefit from the usual resuscitation management of COVID19 , and the experimental group will benefit from losartan and spironolactone treatment in addition to the usual management, according to the study protocol. The number of subjects required has been calculated and 45 patients for each group, for a total of 90 patients.

The SOFA score at D7 will be compared between the "experimental" versus "control" groups using a mean comparison method. The comparison of this criterion and all secondary criteria of judgments between the 2 groups will be performed using a Student or Mann-Whitney test based on the normality of the distribution. The significance threshold will be set at 0.05. No intermediate analysis is scheduled. The analysis will be blinded.

The main expected outcome is an improved prognosis with a decrease in the SOFA severity score at 7 days in resuscitation patients, resulting in an improvement in organ failure. The expected secondary results will be to show the interest of ARA2/Spironolactone treatment on oxygenation based on the PaO2/FiO2 ratio, mechanical ventilation duration and mortality.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is a current pandemic infection caused by an RNA virus called Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2). Severe forms of COVID-19 are most often responsible for isolated respiratory failure in the form of acute respiratory distress syndrome (ARDS), which accounts for most of the mortality. Angiotensin converting enzyme 2 (ACE2) has been shown to be a co-receptor for the entry of SARS-CoV-2 into cells and is likely to play a prolonged role in the pathogenesis of COVID-19. ACE2 and angiotensin (1-7) have been shown to be protective in a number of different lung lesion models. In a mouse model of acidic lung injury, negative regulation of ACE2 by COVID, the SARS virus responsible for the 2003 SARS outbreak, worsened the lung injury which was improved by treatment with ARBs.

We believe that blocking the first RAS pathway at the end of the chain on the AT1r angiotensin 2 receptor may prevent the initiation of this chain reaction and limit decompensation secondary to the disruption of the equilibrium of the renin-angiotensin system. We have several molecules that block the AT1r angiotensin-2 receptor (ARBs) as well as a molecule that blocks the secretion of aldosterone (spironolactone). The main objective is to demonstrate the value of losartan and spironolactone therapy in the regulation of the renin-angiotensin system in improving the prognosis of patients infected with COVID-19 and suffering from acute respiratory distress syndrome.

This is a prospective, multicenter, randomized, open-label, controlled, therapeutic trial studying two parallel groups. The population included in this study is any major patient in acute respiratory distress hospitalized in intensive care requiring oxygen support of at least 6L/min and suffering from a PCR-confirmed SARS-cov2 infection. The control group will benefit from the usual resuscitation management of COVID19 , and the experimental group will benefit from losartan and spironolactone treatment in addition to the usual management, according to the study protocol. The number of subjects required has been calculated and 45 patients for each group, for a total of 90 patients.

The SOFA score at D7 will be compared between the "experimental" versus "control" groups using a mean comparison method. The comparison of this criterion and all secondary criteria of judgments between the 2 groups will be performed using a Student or Mann-Whitney test based on the normality of the distribution. The significance threshold will be set at 0.05. No intermediate analysis is scheduled. The analysis will be blinded.

The main expected outcome is an improved prognosis with a decrease in the SOFA severity score at 7 days in resuscitation patients, resulting in an improvement in organ failure. The expected secondary results will be to show the interest of ARA2/Spironolactone treatment on oxygenation based on the PaO2/FiO2 ratio, mechanical ventilation duration and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with respiratory distress requiring oxygen support of 6 liters per minute or more.
* News-Score greater than 6 PCR SARS-CoV-2 positive in a pharyngeal or respiratory specimen,
* Informed Consent

Exclusion Criteria:

* Minor patient,
* Patient deprived of liberty,
* Refusal of the patient to participate in the study,
* Patient for whom measures of therapeutic limitation have been issued justifying the absence of recourse to mechanical ventilation,
* Patient of 80 years or older,
* Pregnant or breastfeeding woman,
* Patient with prior treatment with ARA2 or ACE inhibitors,
* Hypotension justifying treatment with norepinephrine,
* Acute renal failure with a clearance of less than 60ml/min,
* Severe liver failure.
* Intolerance or contraindication to losartan or spironolactone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
SOFA score | 7 days (J7)
  Organ failures will be assessed on the SOFA score on day 7 post-inclusion.

SECONDARY OUTCOMES:
Pa02/Fi02 | day 3; day 7; day 14; day 21 and day 28
  Oxygenation will be assessed using the PaO2/FiO2 ratio on the 3rd, 7th, 14th, 21st, 28th day after inclusion
Duration of mechanical ventilation | 28 days
  The duration of mechanical ventilation will be evaluated by the number of days of ventilation, the number of days without ventilation between inclusion and death or D28
Death | 28 days
  Mortality will be measured by: mortality at D28, hospital mortality, ICU mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No